CLINICAL TRIAL: NCT02126982
Title: Comparative Study of Clinical Efficacy and Safety of Different Clopidogrel Salts in Patients With Cardiovascular Disease. A Multi-center Non-interventional Clinical Trial.
Brief Title: Salts of Clopidogrel: Investigation to ENsure Clinical Equivalence
Acronym: SCIENCE
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Collaborators: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Alexandros Tselepis, Atherothrombosis Research Centre, University of Ioannina
Other Study IDs: 2012-Clo-U-Io-01
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease; Ischemic Stroke; Peripheral Artery Disease; Carotid Artery Disease; Atrial Fibrillation
Keywords: clopidogrel besylate; clopidogrel hydrogen sulfate; Generic clopidogrel; Coronary Artery Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Ischemic Stroke; Peripheral Arterial Disease; Carotid Artery Diseases; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clopidogrel hydrogen sulfate (CHS): Clopidogrel hydrogen sulfate, 75 mg / day
- Clopidogrel Besylate (CB): Clopidogrel Besylate , 75 mg / day

SUMMARY:
Clopidogrel besylate (CB) is not differentiated relative to the orignal clopidogrel hydrogen sulfate (CHS) in the pharmacokinetics and in antiplatelet potency in healthy volunteers. In addition,CB exhibits similar pharmacodynamic properties compared to CHS in patients with a history of acute coronary syndrome (ACS) and in patients with ACS undergoing percutaneous coronary intervention (PCI). However, there is a lack of data on the clinical efficacy and safety of this salt to the original salt in patients with cardiovascular disease. The aim of this study is to investigate the clinical efficacy and safety of CB in relation to that of CHS in patients eligible to receive clopidogrel.

DETAILED DESCRIPTION:
It is now well documented that platelets play an important role in the pathogenesis of acute coronary syndromes. This phenomenon has significantly strengthened the position of antiplatelet drugs in treatment, and prevention of these syndromes. In terms of administration, antiplatelet drugs are divided into two categories, the oral and intravenous medications. Of these, oral medications are the choice for long-term or prophylactic treatment of patients with acute coronary syndrome. Among them, is clopidogrel, which together with aspirin is now the cornerstone of antiplatelet therapy. Indeed, clopidogrel is a widely used antiplatelet drug. It is second in sales worldwide after atorvastatin and has been prescribed to more than 100 million patients worldwide. Clopidogrel can be used as monotherapy or in combination with aspirin. The efficacy in reducing ischemic events in patients with ACS has been shown in more than 15 major clinical studies involving more than 200,000 patients. These studies also proved the safety of clopidogrel to the bleeding complications (only 1-2% per year).Clopidogrel is a second generation thienopyridine that inhibits the binding of ADP to purinergic receptors of platelet membrane. The ADP activates platelets through different receptors coupled to G-proteins. The main receptor for platelet activation by ADP is P2Y12, associated with the adenyl cyclase and cause deactivation of the resulting reduction in the levels of c-AMP. The identification of this receptor led to the complete elucidation of the mechanism of action of clopidogrel, which proved to be an irreversible antagonist P2Y12.

Clopidogrel is a prodrug that, once granted, is absorbed in the intestine by a process in which an important role is played by the protein carrier ABCB1/MDR1. Then clopidogrel is converted in the liver to the pharmacologically active metabolite by the action of cytochrome P450 (CYP450) and mainly isoform CYP2C19 and isoforms CYP3A4, CYP3A5, CYP1A2, CYP2B6 and CYP2C9. It should be noted that 85% of clopidogrel absorbed, hydrolyzed by esterases in the intestinal mucosa and blood to form biologically inactive products while only 15% of the administered drug is converted to its active metabolite, which is a potent, irreversible, selective inhibitor of receptor P2Y12 ADP resulting in the inhibition of the activation of receptor GPIIb / IIIa and thereby preventing platelet aggregation.

Currently, clopidogrel generic forms are available in the market. Indeed, in 2010 and after 10 years of circulation of the original formulation (clopidogrel bisulfate) under the trade names Plavix or Iscover, released new generic formulations of clopidogrel (generic) due to expiration of the period of exclusive marketing using the original formulation. Main difference of generic forms of clopidogrel to the original formulation (clopidogrel bisulfate) is pharmacochemical recommendation salt of clopidogrel, which in the case of generic formulations is benzenesulfonic (besylate) or hydrochloride salt. Generic formulations of clopidogrel have received marketing approval from the health authorities of the European Union. Bioequivalence comparative studies of clopidogrel generic formulations in healthy volunteers for generic clopidogrel bisulfate, clopidogrel besylate and clopidogrel hydrochloride have proven same pharmacodynamic and pharmacokinetic profile. Considering the wide variability of platelet response to clopidogrel treatment and the high incidence of atherothrombotic events in clopidogrel hyporesponsive patients, studies comparing the pharmacodynamic properties of various generic clopidogrel formulations with those of original clopidogrel bisulfate in CAD patients are essential.

Therefore, given the numerous generic clopidogrel salts that are commercially available today, it is of importance to note that any clinical data or research results arising from the use of these formulations in patients with cardiovascular disease should be related to the specific product used and not generally to the generic clopidogrel.

Our group has performed two prospective pharmacodynamic studies comparing the antiplatelet effectiveness of clopidogrel besylate with that of clopidogrel bisulfate in patients with a history of an ACS, and in ACS patients undergoing PCI. In both studies we showed pharmacodynamic bioequivalence in all platelet function tests performed.

There is a strong need of conducting further clinical studies with adequate number of patients with each clopidogrel generic formulation commercially available in order to confirm its therapeutic equivalence with the innovator product.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* age >18 years
* age <85 years
* Patients with an ACS with or without percutaneous coronary intervention, stable CAD, history of an ischemic stroke/TIA, PAD, carotid artery disease or atrial fibrillation
* agree on study participation
* will comply with all required study procedures

Exclusion Criteria:

* >85 years
* <18 years

Patients with

* hypersensitivity reaction or contraindication to clopidogrel,
* active bleeding or history of severe bleeding (peptic ulcer, trauma or intracranial hemorrhage),
* blood coagulation disorders,
* uncontrolled severe hypertension,
* history of drug or alcohol abuse,
* pregnancy or breastfeeding,
* liver disease
* chronic kidney disease,
* malignancy,
* disagree on study participation,
* evidence for poor compliance with all required study procedures

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suitable for the study will be every patient eligible to receive clopidogrel based on the international guidelines. In particular, in the study will participate patients with an acute coronary syndrome (ACS) or having a stable coronary artery disease (CAD). Patients who have experienced an acute ischemic stroke or a transient ischemic attack (TIA) during the previous 6 months or having a history of peripheral artery disease (PAD) or carotid artery disease, will be also eligible for enrollment. Finally, patients with atrial fibrillation (AF) who will refuse or will not be eligible to use of any oral anticoagulant will be included in the study. The study will include at least 1,500 patients (at least 750 will receive clopidogrel hydrogen sulfate and at least 750 clopidogrel besylate).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy End Point | 12 months
  Composite of death from vascular causes (cardiovascular causes or cerebrovascular causes), MI, or stroke for the entire follow-up period.

SECONDARY OUTCOMES:
Secondary Efficacy End Point | up to 6 and 12 months
  Composite of death from any cause, MI, or stroke (ischemic or hemorrhagic), stent thrombosis and PCI during the entire follow-up period

OTHER OUTCOMES:
Primary Safety End Point | up to 6 and 12 months
  The rate of bleeding events as defined by Bleeding Academic Research Consortium (BARC) criteria
Secondary Safety End Point | up to 6 and 12 months
  Urticaria, temporary or permanent interruption of clopidogrel due to urticaria, temporary interruption due to surgery, dental procedures, patient's desire or bleeding, transient thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Tselepis, MD, PhD Professor, Study Chair — University of Ioannina
Locations (1):
- Atherothrombosis Research Centre / Laboratory of Biochemistry, University of Ioannina, Ioannina, Epirus, Greece

REFERENCES:
- [Background] Davi G, Patrono C. Platelet activation and atherothrombosis. N Engl J Med. 2007 Dec 13;357(24):2482-94. doi: 10.1056/NEJMra071014. No abstract available. PMID 18077812
- [Background] Papathanasiou AI, Goudevenos JA, Mikhailidis DP, Tselepis AD. Acute and long-term antiplatelet therapy. Drugs Today (Barc). 2008 May;44(5):331-52. doi: 10.1358/dot.2008.44.5.1215717. PMID 18548136
- [Background] Antithrombotic Trialists' Collaboration. BMJ 2002;324;71-86
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Serebruany VL, Malinin AI, Jerome SD, Lowry DR, Morgan AW, Sane DC, Tanguay JF, Steinhubl SR, O'connor CM. Effects of clopidogrel and aspirin combination versus aspirin alone on platelet aggregation and major receptor expression in patients with heart failure: the Plavix Use for Treatment Of Congestive Heart Failure (PLUTO-CHF) trial. Am Heart J. 2003 Oct;146(4):713-20. doi: 10.1016/S0002-8703(03)00260-6. PMID 14564328
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] Sabatine MS, Cannon CP, Gibson CM, Lopez-Sendon JL, Montalescot G, Theroux P, Claeys MJ, Cools F, Hill KA, Skene AM, McCabe CH, Braunwald E; CLARITY-TIMI 28 Investigators. Addition of clopidogrel to aspirin and fibrinolytic therapy for myocardial infarction with ST-segment elevation. N Engl J Med. 2005 Mar 24;352(12):1179-89. doi: 10.1056/NEJMoa050522. Epub 2005 Mar 9. PMID 15758000
- [Background] Weber AA, Reimann S, Schror K. Specific inhibition of ADP-induced platelet aggregation by clopidogrel in vitro. Br J Pharmacol. 1999 Jan;126(2):415-20. doi: 10.1038/sj.bjp.0702276. PMID 10077233
- [Background] Gachet C. ADP receptors of platelets and their inhibition. Thromb Haemost. 2001 Jul;86(1):222-32. PMID 11487010
- [Background] Lins R, Broekhuysen J, Necciari J, Deroubaix X. Pharmacokinetic profile of 14C-labeled clopidogrel. Semin Thromb Hemost. 1999;25 Suppl 2:29-33. PMID 10440420
- [Background] Gurbel PA, Antonino MJ, Tantry US. Recent developments in clopidogrel pharmacology and their relation to clinical outcomes. Expert Opin Drug Metab Toxicol. 2009 Aug;5(8):989-1004. doi: 10.1517/17425250903107772. PMID 19575629
- [Background] Schwarz UR, Geiger J, Walter U, Eigenthaler M. Flow cytometry analysis of intracellular VASP phosphorylation for the assessment of activating and inhibitory signal transduction pathways in human platelets--definition and detection of ticlopidine/clopidogrel effects. Thromb Haemost. 1999 Sep;82(3):1145-52. PMID 10494779
- [Background] Darius H, Münzel T, Huber K, Sultan E, Walter U. J Kardiol 2009; 16: 412-6.
- [Background] Kim SD, Kang W, Lee HW, Park DJ, Ahn JH, Kim MJ, Kim EY, Kim SW, Nam HS, Na HJ, Yoon YR. Bioequivalence and tolerability of two clopidogrel salt preparations, besylate and bisulfate: a randomized, open-label, crossover study in healthy Korean male subjects. Clin Ther. 2009 Apr;31(4):793-803. doi: 10.1016/j.clinthera.2009.04.017. PMID 19446152
- [Background] Neubauer H, Kruger JC, Lask S, Endres HG, Pepinghege F, Engelhardt A, Bulut D, Mugge A. Comparing the antiplatelet effect of clopidogrel hydrogensulfate and clopidogrel besylate: a crossover study. Clin Res Cardiol. 2009 Sep;98(9):533-40. doi: 10.1007/s00392-009-0033-1. Epub 2009 Jun 6. PMID 19504141
- [Background] Borsiczky B, Sarszegi Z, Konyi A, Szabados S, Gaszner B. The effect of clopidogrel besylate and clopidogrel hydrogensulfate on platelet aggregation in patients with coronary artery disease: a retrospective study. Thromb Res. 2012 Jun;129(6):700-3. doi: 10.1016/j.thromres.2011.08.013. Epub 2011 Sep 15. PMID 21924759
- [Background] Tsoumani ME, Kalantzi KI, Dimitriou AA, Ntalas IV, Goudevenos IA, Tselepis AD. Antiplatelet efficacy of long-term treatment with clopidogrel besylate in patients with a history of acute coronary syndrome: comparison with clopidogrel hydrogen sulfate. Angiology. 2012 Oct;63(7):547-51. doi: 10.1177/0003319711427697. Epub 2011 Dec 5. PMID 22144668
- [Background] Tsoumani ME, Kalantzi KI, Dimitriou AA, Ntalas IV, Goudevenos IA, Tselepis AD. Effect of clopidogrel besylate on platelet reactivity in patients with acute coronary syndromes. Comparison with clopidogrel hydrogen sulfate. Expert Opin Pharmacother. 2012 Feb;13(2):149-58. doi: 10.1517/14656566.2012.644536. Epub 2011 Dec 21. PMID 22188544
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Derived] Ntalas IV, Kalantzi KI, Tsoumani ME, Bourdakis A, Charmpas C, Christogiannis Z, Dimoulis N, Draganigos A, Efthimiadis I, Giannakoulas G, Giatrakos I, Giogiakas V, Goumas G, Hatziathanasiou G, Kazakos E, Kipouridis N, Konstantinou S, Milionis H, Nikolopoulos D, Peltekis L, Prokopakis N, Sinteles I, Stroumbis C, Terzoudi K, Thoma M, Tsilias K, Vakalis I, Vardakis K, Vasilakopoulos V, Vemmos K, Voukelatou M, Xaraktsis I, Panagiotakos DB, Goudevenos JA, Tselepis AD. Salts of Clopidogrel: Investigation to Ensure Clinical Equivalence: A 12-Month Randomized Clinical Trial. J Cardiovasc Pharmacol Ther. 2016 Nov;21(6):516-525. doi: 10.1177/1074248416644343. Epub 2016 Apr 14. PMID 27081185
- [Derived] Ntalas IV, Kalantzi KI, Tsoumani ME, Vakalis JN, Vasilakopoulos V, Vardakis K, Vemmos KN, Voukelatou M, Giannakoulas G, Giatrakos I, Giogiakas V, Goumas G, Dimoulis N, Draganigos A, Efthimiadis I, Thoma M, Kazakos E, Kipouridis N, Konstantinou S, Bourdakis A, Nikolopoulos D, Peltekis L, Prokopakis N, Sinteles I, Stroumbis CS, Terzoudi K, Tsilias K, Xaraktsis I, Charmpas C, Hatziathanasiou G, Christogiannis Z, Panagiotakos DB, Goudevenos JA, Tselepis AD. Generic Clopidogrel Besylate in the Secondary Prevention of Atherothrombotic Events: A 6-month Follow-up of a Randomised Clinical Trial. Curr Vasc Pharmacol. 2015;13(6):809-18. doi: 10.2174/1570161113666150316220515. PMID 25782408